CLINICAL TRIAL: NCT07157072
Title: Effect of Innominate Rigid Taping on Gait and Balance in Patients With Unilateral Chronic Ankle Instability Associated With Pelvic Torsion
Brief Title: Effect of Pelvic Rigid Taping on Gait and Balance in Chronic Ankle Instability Patients With Pelvic Torsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Saeed Abdul Haleem, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/005797
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: Gait; Balance; Pelvic torsion; Rigid taping; Chronic ankle instability

STUDY DESIGN:
Intervention Model Description: A single group with repeated measurement design was used to evaluate the effect of rigid taping on gait and balance over four time points: pre-intervention, immediately,1 week, and 2 weeks post- intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental single group (Experimental): Single group who received application of corrective rigid taping for a period of 2 weeks to correct pelvic torsion and examine the effect of that correction on gait and balance
  Interventions: Other: Corrective rigid taping

INTERVENTIONS:
Other: Corrective rigid taping — Rigid taping used to correct pelvic torsion in patients with CAI

SUMMARY:
Ankle sprain is one of the most common musculoskeletal injuries, with a high incidence among physically active individuals. acute ankle sprains associated with the development of chronic ankle instability (CAI) which has been found to affect the whole lower quarter kinetic chain. This chronicity decrease the physical activity level and quality of life, All these consequences cost the patients physically, emotionally, socially and financially. Purpose: To investigate the effect of corrected pelvic torsion using rigid taping on gait parameters and balance in patients with unilateral CAI associated with pelvic torsion.

DETAILED DESCRIPTION:
Background: Ankle sprain is one of the most common musculoskeletal injuries, with a high incidence among physically active individuals. acute ankle sprains associated with the development of chronic ankle instability (CAI) which has been found to affect the whole lower quarter kinetic chain. This chronicity decrease the physical activity level and quality of life, All these consequences cost the patients physically, emotionally, socially and financially. Purpose: To investigate the effect of corrected pelvic torsion using rigid taping on gait parameters and balance in patients with unilateral CAI associated with pelvic torsion. Materials and Methods: 22 subjects from both genders were assessed for the presence of unilateral CAI associated with pelvic torsion , gait and balance were assessed using teckscan walkway assessment system and biodex balance system then rigid tape applied to the anteriorly tilted innominate then gait and balance reassessed again immediately after taping ,after one week and after two weeks.

ELIGIBILITY:
Inculsion criteria :

1. history of at least one significant ankle sprain (the initial sprain must have occurred at least 12 months prior to study enrollment and the most recent injury must have occurred more than 3 months prior to study enrollment.
2. Participants should report at least 2 episodes of giving way in the last 6 month.
3. Self-reported ankle instability using CAIT should be >24 .
4. the presence of pelvic torsion must be present and confirmed using the PALM-Meter .

Exclusion criteria:

1. Individuals with bilateral lateral anklesprain.
2. Those with low back pain that required medical or surgical intervention.
3. Those with a history of spine, pelvis, and lower extremity injury, fracture, or surgery.
4. patients with trunk asymmetry angle of more than 7º and leg length discrepancy of more than 0.5 cm(19), those with skin diseases or sensitivity to rigid

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Overall Stability Index measured by Biodex Balance System | Baseline, immediately post-intervention(Day 1), one week post-intervention(week 1), two weeks post-intervention(week 2)
  Change in overall stability index using the Biodex Balance System
Anterior/Posterior Stability Index measured by Biodex Balance System | Baseline, immediately post-intervention (Day1), 1 week post-intervention, 2 weeks post intervention.
  Change in anterior/posterior stability index using the Biodex Balance System
Medial/Lateral Stability Index measured by Biodex Balance System | Baseline, immediately post-intervention (Day1), 1 week post-intervention, 2 weeks post intervention.
  Change in medial/lateral stability index using the Biodex Balance System
Maximum peak plantar pressure assessed using Tekscan walkway system. | Baseline, immediately post-intervention (Day1), 1 week post-intervention, 2 weeks post-intervention.
  Maximum peak pressure(N/cm²) during walking as measured using the Tekscan walkway system. This represents the highest pressure recorded under the foot during gait.
Walking Velocity | Baseline, immediately post-intervention (Day1), 1 week post-intervention, 2 weeks post-intervention
  Average walking speed (m/s) during gait assessment using the Tekscan walkway system. Calculated as distance traveled divided by time taken.
Cadence | Baseline, immediately post-intervention(Day 1), 1 week post-intervention, 2 weeks post- intervention.
  Number of steps taken per minute (steps/min) during walking assessment using the Tekscan walkway system.
Step length | Baseline, immediately post-intervention (Day1), 1 week post-intervention, 2 weeks post-intervention.
  Average distance(m) between successive heel contacts of opposite feet during walking, measured using the Tekscan walkway system.

CONTACTS AND LOCATIONS:
Overall Officials: Enass F Youssef, Professor, Study Chair — Cairo University
Locations (1):
- Faculty of physical therapy, mti university, Cairo, El Mokkatem, Egypt

IPD SHARING:
Plan to Share IPD: No